CLINICAL TRIAL: NCT02770937
Title: A Prospective Randomized Controlled Trial Comparing Virtual Reality Simulation Training and Box Trainer on the Acquisition of Laparoscopic Suturing Skills
Brief Title: Simulator Versus Box Trainer on Laparoscopic Suturing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HKUCTR-1920
Record Dates: First submitted 2016-05-03; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Simulation Training, Laparoscopy
Keywords: laparoscopy, simulator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Virtual reality simulator (Active Comparator): The virtual reality simulator group will receive a maximum of 4 hours of training (2 sessions, 2 hours each) using the Simbionix simulator on laparoscopic suturing.
  Interventions: Other: Virtual reality simulator; Device: Simbionix
- Box trainer (Active Comparator): The box trainer group will receive a maximum of 4 hours of training (2 sessions, 2 hours each) using the Simbionix simulator on box trainer.
  Interventions: Other: Box trainer; Device: Simbionix
- Control (No Intervention): The control group will not receive further training.

INTERVENTIONS:
Other: Virtual reality simulator — The virtual reality simulator group will receive a maximum of 4 hours of training (2 sessions, 2 hours each) using the Simbionix simulator on laparoscopic suturing.
  Arms: Virtual reality simulator
Other: Box trainer — The box trainer group will receive a maximum of 4 hours of training (2 sessions, 2 hours each) on a box trainer.
  Arms: Box trainer
Device: Simbionix
  Arms: Box trainer; Virtual reality simulator

SUMMARY:
This is prospective randomized controlled study to compare the proficiency of novices in acquiring laparoscopic suturing skills following either training in a virtual reality simulator or box trainer.

DETAILED DESCRIPTION:
Participants will be randomized into three groups by computer-generated sequence to the virtual reality simulator, box trainer and control groups. They will be shown a video demonstration and given simple instructions on laparoscopic suturing and intracorporeal knot tying at the beginning of the training. Both the virtual reality simulator and box trainer groups will be allowed a maximum of 4 hours of training (2 sessions of 2 hours each). The participants could terminate training at any time point during the 4-hour if they felt competent to perform the task.The control group will not receive any further training.

They will then be asked to perform laparoscopic suturing (which would involve needle loading and insertion via 2 pre-marked circles, and knot tying which includes at least 2 single throws) on a box trainer. Participants will be asked to complete a modified GOALS questionnaire at the end (which will take around 5 minutes) to evaluate their experiences and assess their own proficiency. The procedure will also be recorded (with a number identifying the participant only) and assessment will be performed when the study is completed by 2 experienced laparoscopic gynecologists blinded to the participants who will review the recorded procedure. The time to complete each task, total procedural time and proficiency will be assessed, which will be compared against the participants' own evaluation.

ELIGIBILITY:
Inclusion Criteria:

All trainees and interns working in the Department of Obstetrics and Gynecology who have (i) no laparoscopic experience or (ii) laparoscopic experience but no laparoscopic suturing experience, will be invited to participate in the study.

* Older than the age of legal consent (i.e. 18 years old)
* Willing and able to participate after the study has been explained

Exclusion Criteria:

- Cannot understand English, Cantonese or Putonghua

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The time to complete task | within 10 days after completion of training
Surgeon's preference (modified GOALS questionnaire score) | Within 10 days after completion of training
Objective score | Within 3 months after completion of training and assessment
  Scored by 2 experienced gynecological laparoscopists

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No